CLINICAL TRIAL: NCT06076304
Title: Nasal Steroids, Irrigation, Oral Antibiotics, and Subgroup Targeting for Effective Management of Sinusitis
Acronym: NOSES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Merenstein (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Medstar Health Research Institute (Other); Penn State College of Medicine (Unknown); University of Washington (Other); Virginia Commonwealth University (Other); University of California, Los Angeles (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Daniel Merenstein, Director of Research Programs, Department of Family Medicine, Principal Investigator, Professor, Georgetown University
Organization: Georgetown University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLACER-2021C3-24476; 23-02-622 (Other: IRB)
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sinus Infection; Acute Sinusitis
Keywords: sinusitis; antibiotics; intranasal corticosteroids; saline nasal irrigation; comparative effectiveness
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination; Budesonide; C-Reactive Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- antibiotic (Active Comparator): amoxicillin/clavulanate
  Interventions: Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet; Other: C-reactive protein
- placebo antibiotic (Placebo Comparator): placebo antibiotic, amoxicillin/clavulanate
  Interventions: Drug: Placebo; Other: C-reactive protein
- antibiotic plus intranasal corticosteroid (Active Comparator): amoxicillin/clavulanate plus budesonide
  Interventions: Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet; Drug: Budesonide nasal spray; Other: C-reactive protein
- placebo antibiotic plus intranasal corticosteroid (Other): placebo antibiotic plus budesonide
  Interventions: Drug: Placebo; Drug: Budesonide nasal spray; Other: C-reactive protein

INTERVENTIONS:
Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet — Amoxicillin/clavulanate, oral, 875mg/125mg twice daily for 7 days
  Other Names: Augmentin
  Arms: antibiotic; antibiotic plus intranasal corticosteroid
Drug: Placebo — Placebo for amoxicillin/clavulanate, oral, twice daily for 7 days
  Other Names: Inactive; Control
  Arms: placebo antibiotic; placebo antibiotic plus intranasal corticosteroid
Drug: Budesonide nasal spray — Budesonide nasal spray, 32 mcg per spray, 2 sprays per nostril, once per day
  Other Names: Rhinocort
  Arms: antibiotic plus intranasal corticosteroid; placebo antibiotic plus intranasal corticosteroid
Other: C-reactive protein — Measurement of C-reactive protein level in capillary blood
  Other Names: CRP

SUMMARY:
Sinus infections are sometimes treated with oral antibiotics or nasal steroid sprays, while some patients get better on their own. Some patients may wait a few days or use common over-the-counter remedies to see if their symptoms improve without further treatment. Sometimes this is enough to help patients wait a few days to see if their infection clears up without needing to use antibiotics or nasal steroid sprays. The overall goal of this clinical trial to see which specific groups of patients benefit more from which intervention or combination of intervention, and which improve with supportive care alone.

DETAILED DESCRIPTION:
One in seven adults are diagnosed with acute sinus infections (also known as rhinosinusitis or ARS) every year in the United States, for an annual total of 30 million office visits. Most acute sinus infections seen in outpatient setting are caused by viral infection, but antibiotics are prescribed in over 70% of these visits. The overarching goal is to improve outcomes for patients with ARS by understanding which subgroups are most likely to benefit from antibiotics, supportive care, watchful waiting, intranasal corticosteroids (INCS), or a combination of treatments.

To assess the comparative effectiveness of the treatments, a large, pragmatic, randomized controlled trial, will be conducted in primary and urgent care clinics within six geographical areas. Enrolled adults ages 18-75 years presenting to a clinician with symptoms consistent with ARS will enter the study in one of 2 phases, dependent on the number of days with symptoms. Phase 1 is a pre-randomization, waiting period of 9 or more days, with options for supportive care. Patients who qualify will enter Phase 2 and will be randomly assigned to one of the four arms. All groups will use approved or over-the counter drugs or spray, or a placebo (inactive or dummy pill). Patients will be in Phase 2 for approximately 14 days. All patients will complete a two-minute daily diary and periodic follow-ups about their symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old; AND are experiencing either:
2. "persistent" symptoms or signs compatible with ARS or sinus infection lasting for 1-21 days without any evidence of clinical improvement (Symptoms include facial pain or pressure, facial congestion or fullness, nasal obstruction, nasal discharge, no or reduced sense of smell, fever ≤39°C or 102°F, headache, bad smelling breath, fatigue, ear pain or pressure, and dental pain); OR
3. onset with worsening symptoms or signs characterized by the new onset of fever, headache, or increase in nasal discharge following a typical viral upper respiratory infection (URI) that lasted 5-6 days and were initially improving (''double-sickening'').

Exclusion Criteria:

* allergy or intolerance to penicillin
* received systemic antibiotic therapy in the past 4 weeks
* prior sinus surgery (cosmetic surgery, such as rhinoplasty, septal deviation, etc. are not exclusionary)
* complications of sinusitis (facial edema (swelling), cellulitis), or orbital, meningeal or cerebral signs)
* health care clinician determined IV (intravenous) antibiotics or hospital admission are required
* pregnancy or breastfeeding
* presence of a comorbidity or medication that may impair a patient's immune response as determined by a health care clinician
* hospitalization in past 5 days
* unable or unwilling to provide informed consent or comply with study protocol requirements
* fever >39°C or 102°F today
* taking intranasal corticosteroids (INCS) regularly in the past two weeks and unwilling to stop its use while in the study; OR
* previously enrolled or participated in the feasibility phase or this stage of study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3720 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms | day 1 and 3 days post-randomization
  Improvement of symptoms will be assessed using the Modified Sino-Nasal Outcome Test (mSNOT-16), a disease-specific quality of life questionnaire. Sixteen sinus symptoms are self-assessed on a 0-3 point scale, with 0=No Problem, 1=Mild or Slight Problem, 2=Moderate Problem, 3=Severe Problem. Scores will be measured at day 1 and 3 days post-randomization.

SECONDARY OUTCOMES:
Improvement of symptoms | baseline to 14 days post-randomization
  Improvement of symptoms will be assessed using the Modified Sino-Nasal Outcome Test (mSNOT-16), a disease-specific quality of life questionnaire. Sixteen sinus symptoms are self-assessed on a 0-3 point scale, with 0=No Problem, 1=Mild or Slight Problem, 2=Moderate Problem, 3=Severe Problem. Scores will be measured at daily from baseline until 14 days post-randomization.
Work Productivity and Activity Impairment Questionnaire | Baseline, 9 days of symptoms, and 1, 7, and 14 days post-randomization
  The Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI: SHP) 2.0 is a 6-question self-reported questionnaire on the effects of sinus symptoms on the amount of absenteeism, presenteeism, work impairment, and daily activity impairment. WPAI will be assessed at baseline, 9 days of symptoms is reached, and 1, 7, and 14 days post-randomization.
Global Rating of Improvement | Baseline, 9 days of symptoms, and 3, 7, and 14 days post-randomization
  Self-assessment of current sinus symptoms at each follow-up interview using a 6-point categorical scale (1=no symptoms, 2=a lot better, 3=a little better, 4=the same, 5=a little worse, or 6=a lot worse). Scores will be measured at baseline, when 9 days of symptoms is reached, and 3, 7, and 14 days post-randomization.
Symptomatic care | Baseline to 14 days post-randomization
  Number of patients reporting use of over-the-counter medicines or supplements during the pre- and post-randomization study periods.
Adverse events | Baseline to 14 days post-randomization
  Number of adverse events reported during a follow-up or on the diary during the the pre- and post-randomization study periods. Events are graded form 1-5 using the NCI Common Terminology Criteria for Adverse Events.

OTHER OUTCOMES:
Saline nasal irrigation | Baseline to 14 days post-randomization
  Number of patients reporting use of saline nasal irrigation during the pre- and post-randomization study periods.
Watchful waiting | Baseline to 9 days of symptoms
  Number of patients who experienced improvement or resolution of symptoms during the pre-randomization period (between enrollment and 9 days of symptoms).
Adherence | Days 1-7 post-randomization
  Self-reported adherence to study pill and nasal spray are calculated by [number of doses taken]/[prescribed number of doses] x 100, over the 7-day intervention period.
C-reactive protein (CRP) | Baseline
  Measurement of C-reactive protein (CRP) level in capillary blood
Other signs and symptoms of ARS | Baseline to 14 days post-randomization
  Number of patients who experienced double-sickening, evidence of purulence, change of smell, pain in the teeth, clinician impression/gestalt, facial or nasal congestion or fullness, no or reduced sense of smell, fever ≤39°C or 102°F, bad smelling breath

CONTACTS AND LOCATIONS:
Overall Officials: Dan Merenstein, MD, Principal Investigator — Georgetown University
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No